CLINICAL TRIAL: NCT00594191
Title: Phase IV-II Randomized, Multicenter, Placebo-Controlled Double-Blind Clinical Trial Evaluating the Effects of Continuous Simvastatin Administration on Hepatic and Systemic Hemodynamics in Patients With Cirrhosis.
Brief Title: Efficacy and Safety of Simvastatin in the Treatment of Portal Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Jaime Bosch /Professor of Medicine, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIMV-HTP2003; AEM 03-0434
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Cirrhosis; Portal Hypertension
Keywords: Statins; HMG-CoA reductase inhibitors; Cirrhosis; Portal hypertension; Variceal bleeding
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 20 mg/day p.o., increased to 40 mg/day at day 15 if no safety end-point was met
  Arms: B
Drug: Placebo — Placebo with the same characteristics of the drug and at the same dose
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the effects of continuous simvastatin administration on the hepatic venous pressure gradient (HVPG), as a surrogate marker of prognosis, and its safety in patients with cirrhosis and portal hypertension.

DETAILED DESCRIPTION:
Statins exert beneficial vascular effects independently of cholesterol reduction by improving endothelial dysfunction. In cirrhosis sinusoidal endothelial dysfunction further increases intrahepatic resistance and portal pressure. Previous studies have shown that statins improve hepatic endothelial dysfunction in cirrhosis, suggesting that statins could be an effective therapy for portal hypertension (PHT). This randomized controlled trial evaluated the effects of continuous simvastatin administration on the hepatic venous pressure gradient (HVPG), as a surrogate marker of prognosis, and its safety in patients with cirrhosis and PHT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75.
2. Clinical, analytical, ultrasound or pathological criteria of cirrhosis.
3. Severe sinusoidal portal hypertension (HVPG >12 mmHg)
4. Signed informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Advanced liver disease defined as one of the following: Prothrombin rate <40%, Bilirubin >5 mg/dl, hepatic encephalopathy > grade I or Child-Pugh score >12).
3. Portal vein thrombosis
4. Multinodular hepatocellular carcinoma or single hepatocellular carcinoma > 5 cm.
5. Heart, renal or respiratory failure
6. Previous portal-systemic shunt
7. Treatment with organic nitrates
8. Hypersensitivity to HMG-CoA reductase inhibitors
9. Previous treatment with HMG-CoA reductase inhibitors
10. Treatment with calcium channel blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-03; Primary Completion 2007-04 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Changes in hepatic venous pressure gradient (HVPG) | 4 weeks

SECONDARY OUTCOMES:
Changes in systemic hemodynamics | 4 weeks
Changes in liver function tests | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Bosch, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (3):
- Spain (3):
  - Hepatic Hemodynamic Laboratory. Liver Unit. Hospital Clinic., Barcelona, Barcelona
  - Servicio de Gastroenterología, Hospital Ramón y Cajal, Madrid, Madrid
  - Servicio de Gastroenterología, Hospital Universitario General Gregorio Marañón, Madrid, Madrid